CLINICAL TRIAL: NCT02286219
Title: Phase 1, Multiple Ascending Dose Study of Anti-HER2 FCAB FS102 in HER2 Positive Solid Tumors
Brief Title: Phase 1, Multiple Ascending Dose Study of Anti-HER2 FCAB FS102 in HER2 Positive Solid Tumors (Anti HER2 Fcab)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CA014-001; FS10214100 (Other: F-star Alpha, Ltd)
Record Dates: First submitted 2014-10-31; First posted 2014-11-07 (Estimated); Last update posted 2017-09-18 (Actual); Status verified 2017-09

CONDITIONS: Solid Tumors That Overexpress HER2 (HER2 Positive)
MeSH Terms: interventions — Immunoglobulin G

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- FS102 (Experimental): Dose escalation of either weekly or Q3W of FS102
  Interventions: Drug: FS102

INTERVENTIONS:
Drug: FS102 — Experimental
  Other Names: Fcab, Fc region of full immunoglobulin G, subclass 1 [IgG1]

SUMMARY:
To evaluate the safety, tolerability, dose limiting toxicity (DLT), and maximum tolerated dose (MTD), of FS102(BMS-986186) when administered intravenously (IV) to subjects with relapsed or refractory solid tumors that overexpress HER2 and who have no standard treatment options.

DETAILED DESCRIPTION:
This is a Phase 1, open-label, multiple dose escalation study in subjects with solid tumors that over express HER2.

Subjects with locally un-resectable and/or metastatic solid cancers that over express human epidermal growth factor tyrosine kinase receptor 2 (HER2) by standard clinical pathology criteria and who have no standard treatment options will be enrolled into a series of escalating dose cohorts.

Within each dose cohort, subjects will receive weekly (± 1 day) or less frequent IV (Q3W) infusions of FS102 during an initial 28-day (4-week) DLT observation period. During the DLT observation period, subjects will be assessed for safety, tolerability, dose limiting toxicity, PK, immunogenicity, and clinical disease response. Following assessment by the Investigator, subjects without clinical disease progression and without unacceptable toxicity will be eligible to continue receiving FS102 for up to six 21 (Q3W) to 28-day (weekly) cycles.

Continuation Phase. Subjects who complete six 21-28-day cycles of treatment will be evaluated for entry into an extended Continuation Phase of the study. Subjects will be eligible for continuation if:

* They demonstrate no evidence of disease progression;
* In the opinion of the Investigator they are deemed reasonably likely to continue to benefit from treatment; and
* They have not experienced any toxicity requiring discontinuation. During the Continuation Phase, subjects will continue to receive FS102 at the same dose they were originally assigned, unless modified downward for earlier toxicity. No dose escalation within subjects will be permitted.

Treatment may continue until one of the following criteria applies:

* Disease progression;
* Intervening illness that prevents further administration of treatment;
* Unacceptable adverse events;
* Significant subject non-compliance with protocol;
* Pregnancy;
* Subject decides to withdraw from study;
* General or specific changes in the subject's condition that render the subject unacceptable for further treatment in the judgment of the Investigator; or
* Sponsor decides to end the study.

ELIGIBILITY:
For more information regarding BMS clinical trial participation, please visit www.BMSStudyConnect.com

Inclusion Criteria:

1. Signed written informed consent obtained prior to performing any study procedure, including screening procedures.
2. Men and women ≥ 18-years-old on the day of signing informed consent.
3. Subjects must have histologically or cytologically confirmed solid tumor malignancy that is unresectable/locally advanced and/or metastatic and for which standard curative or palliative measures are not available or are no longer effective (for all subjects, histologic or cytologic proof of malignancy based on prior primary cancer pathology is acceptable).
4. Subjects must have HER2-positive tumors and written clinical pathology report documentation of HER2 status available for Sponsor's Medical Monitor review.

   1. Assessment of HER2 status in subjects with breast cancer should follow the 2013 American Society of Clinical Oncology (ASCO)/College of American Pathologists (CAP) criteria (Wolff et al, 2013) as practicable.
   2. Assessment of HER2 status in subjects with gastric and gastroesophageal junction adenocarcinoma should follow the criteria published by Rüschoff et al (2012) as practicable.
   3. Assessment of HER2 status in subjects with non-breast/non-gastric cancers may follow local institutional criteria. These criteria should be made available to the Sponsor.
   4. All subjects with breast and gastric/gastroesophageal junction cancers should have HER2 testing performed using an assay kit/methodology specifically FDA-approved for their cancer type as practicable.
   5. Subjects for whom the clinical pathology report includes only IHC as 3+ (does not reflex to ISH) may enroll without a written report of ISH determined HER2 copy number, provided the investigative site confirms that archival tissue is available.
5. Subjects with breast cancer must have been treated with at least two FDA-approved anti-HER2 directed therapies (more than two is also permissible), and subjects with gastric and gastroesophageal junction cancers must have been treated with at least one FDA-approved anti-HER2 directed therapy (more than one is also permissible); and all subjects must have refractory or relapsed/progressive disease during or following their last prior anti-HER2 directed therapy.

   1. Subjects enrolling in the study who have non-breast, non-gastric, non-gastroesophageal junction cancers do not require any prior treatment with anti-HER2 therapy if there is no FDA-approved anti-HER2 agent for their specific cancer type, but they must have refractory or relapsed/progressive disease during or following their last prior anti-cancer therapy.
   2. For all subjects, prior post-operative adjuvant administration of anti-HER2 therapy is permissible.
6. Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0-1 and estimated life expectancy ≥ 3 months.
7. Any prior cumulative doxorubicin dose must be ≤ 360 mg/m2; prior cumulative epirubicin dose must be ≤ 720 mg/m2.
8. Adequate organ function as defined below:

   1. Serum aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 2.5 upper limit of normal (ULN); if liver function abnormalities are due to the underlying malignancy, then AST and ALT must be ≤ 5 ULN;
   2. Total serum bilirubin ≤ ULN unless due to Gilbert's Syndrome;
   3. Serum creatinine ≤ 1.25 x ULN; or if serum creatinine > 1.25 ULN, then calculated (Cockcroft-Gault formula, glomerular filtration rate (GFR) ≥ 60 mL/min;
   4. Hemoglobin ≥ 9.0 g/dL and not requiring > 1 unit red blood cell transfusion per month; subjects receiving therapeutic erythropoietin preparations in accordance with the FDA product label are eligible to enroll;
   5. Absolute neutrophil count ≥ 1,500/mm3 (not supported by growth factors in the preceding 21 days);
   6. Platelet count ≥ 100,000/mm3 (without platelet transfusion or growth factor support in the preceding 7 days);
   7. Activated partial thromboplastin time (aPTT) ≤ 1.25 ULN and international normalized ratio (INR) ≤ 1.3 (unless the subject is receiving therapeutic anticoagulants);
   8. Left ventricular ejection fraction (LVEF) determined by 2 dimensional echocardiogram (2D Echo) or multi-gated acquisition scan (MUGA) ≥ 50% or ≥ local institutional lower limit normal (LLN) whichever is higher.
   9. Serum magnesium, calcium, and phosphorus must be within normal reference ranges as per local tests. [If initial screening results are outside of normal reference range, the Investigator may initiate appropriate measures to correct. However administration of FS102 may not proceed until the specified electrolytes have normalized.]
9. Women of childbearing potential (WOCBP) must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of HCG) during screening for eligibility assessments and enrollment and within 24 hours prior to the start of study drug.
10. Women must not be breastfeeding
11. WOCBP must agree to follow instructions for method(s) of contraception for the duration of treatment with study drug FS102 plus 30 days (duration of ovulatory cycle) for a total of 30 days post-treatment completion.
12. Males who are sexually active with WOCBP must agree to follow instructions for method(s) of contraception for the duration of treatment with study drug FS102 plus 90 days (duration of sperm turnover) for a total of 90 days post-treatment completion.
13. Azoospermic males and WOCBP who are continuously not heterosexually active are exempt from contraceptive requirements. However they must still undergo pregnancy testing as described in this section.

Investigators shall counsel WOCBP and male subjects who are sexually active with WOCBP on the importance of pregnancy prevention and the implications of an unexpected pregnancy. Investigators shall advise WOCBP and male subjects who are sexually active with WOCBP on the use of highly effective methods of contraception. Highly effective methods of contraception have a failure rate of < 1% when used consistently and correctly.

At a minimum, subjects must agree to the use of two methods of contraception, with one method being highly effective and the other method being either highly effective or less effective as listed below.

Exclusion Criteria:

1. Primary brain or other central nervous system malignancy.
2. Any history of leptomeningeal metastasis.
3. Active brain metastasis or treatment for brain metastasis within 1 month of scheduled dosing day 1.

   a. Dose of corticosteroid, if any, for brain metastasis must be tolerated in terms of glucose tolerance ≤ Grade 2 (symptomatic; dietary modification or oral agent indicated) and hyperglycemia ≤ Grade 2 (fasting glucose value >160 - 250 mg/dL [> 8.9 - 13.9 mmol/L]).
4. History of second or other primary cancer with the exception of: 1) curatively treated non-melanomatous skin cancer; 2) curatively treated cervical or breast carcinoma in situ; or 3) other primary solid tumor treated with curative intent and no known active disease present and no treatment administered during the last 3 years.
5. Receipt of any investigational treatment within 4 weeks of scheduled dosing day 1.
6. Receipt of cytotoxic chemotherapy within 3 weeks (6 weeks for nitrosoureas and mitomycin C) of scheduled dosing day 1.
7. Receipt of radiation therapy within 3 weeks of scheduled dosing day 1, unless the radiation comprised a limited field to non-visceral structures (eg, a limb bone metastasis).
8. Receipt of treatment with immunotherapy (including interferons, interleukins, immunoconjugates), biological therapies (including monoclonal antibodies or other engineered proteins), targeted small molecules (including but not limited to kinase inhibitors), hormonal therapies (except for gonadotropin releasing hormone agonists/antagonists for prostate cancer which may be continued while on study) within 3 weeks of scheduled dosing day 1.
9. Receipt of trastuzumab, pertuzumab, or ado-trastuzumab emtansine within 4 weeks of scheduled dosing day 1.
10. Receipt of lapatinib within 7 days of scheduled dosing day 1.
11. Is concurrently enrolled in another therapeutic clinical trial involving ongoing therapy with any investigational or marketed product or placebo.
12. Exclusionary concurrent medical conditions:

    1. Hypertension which is not controlled to systolic < 160 mm Hg and diastolic < 90 mm Hg;
    2. Myocardial infarction, unstable angina, coronary artery bypass graft, coronary artery angioplasty or stent placement within 12 months before scheduled dosing day 1;
    3. History of congestive heart failure;
    4. History of absolute decrease in LVEF of ≥ 16 absolute percentage points, or ≥ 10 absolute percentage points and crossing from > LLN to < LLN on prior anti-HER2 therapy, even if asymptomatic and the LVEF decrease recovered;
    5. Abnormal 12-lead electrocardiogram (ECG) judged to be clinically significant by the Investigator;
    6. Hemorrhagic, embolic, or thrombotic stroke within 6 months of scheduled dosing day 1;
    7. Prior bone marrow or stem cell transplant;
    8. Previously known infection with human immunodeficiency virus (HIV); or, hepatitis B or C requiring treatment;
    9. Any active infection requiring the use of parenteral anti-microbial agents or that is > Grade 2;
    10. Non-malignant interstitial lung disease;
    11. Dyspnea of any cause requiring supplemental oxygen therapy;
    12. Significant traumatic injury or major surgery (major surgery means opening of a body cavity, eg, thoracotomy, laparotomy, laparoscopic organ resection, and major orthopedic procedures, eg, joint replacement, open reduction and internal fixation) within 21 days of scheduled dosing day 1;
    13. Any other acute or chronic medical or psychiatric condition (including alcohol and illicit substance abuse) or laboratory abnormality that could increase the risk associated with study participation or could interfere with the interpretation of the study results and, in the judgment of the Investigator or Medical Monitor, would render the subject inappropriate for participation in the study.
13. Has not recovered from the adverse effects of previous anti-cancer treatments to pre-treatment baseline or Grade 1, except for alopecia, anemia (hemoglobin must meet the present study inclusion criterion), and peripheral neuropathy (which must have recovered to ≤ Grade 2).
14. Hypersensitivity/infusion reaction to monoclonal antibodies, other therapeutic proteins, or allergy to any component/excipient of FS102 finished drug product (arginine, glycine, phosphoric acid, or polysorbate 80) and the reaction could not be controlled or prevented on subsequent infusion with standard therapies such as anti-histamines, 5-HT3 antagonists, or corticosteroids.
15. Subjects who are pregnant or breast feeding.
16. Subjects who are unable or unwilling to comply with all study requirements for clinical visits, examinations, tests, and procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2014-11-04 (Actual); Primary Completion 2017-06-08 (Actual); Study Completion 2017-06-08 (Actual)

PRIMARY OUTCOMES:
Adverse events as assessed by NCI Common Toxicity Criteria for Adverse Events CTCAE v3.0 | 1 year

SECONDARY OUTCOMES:
Clinical benefit as assessed by objective response rate | 1 year
PK profile as assessed by drug levels | 1 year
Adverse events as assessed by immune response to drug | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (6):
- United States (5):
  - Anthony El-Khoueiry, Md, Los Angeles, California
  - MedStar Georgetown University Hospital, Washington D.C., District of Columbia
  - The West Clinic, Memphis, Tennessee
  - Southwest Texas Addiction Research And Tech (Start) Center, San Antonio, Texas
  - University of Washington, Seattle, Washington
- The Ottawa Hospital Cancer Centre, Ottawa, Ontario, Canada

REFERENCES:
- See also: BMS Clinical Trial Patient Recruiting — http://bms.com/studyconnect/Pages/home.aspx
- See also: Investigator Inquiry Form — http://www.bms.com/clinical_trials/Pages/Investigator_inquiry_form.aspx